CLINICAL TRIAL: NCT05804383
Title: A Phase 1B Multiple Ascending Dose Study of The Safety and Tolerability of BMS-984923 in Healthy Older Adults and Patients With Alzheimer's Disease
Brief Title: A Multiple Ascending Dose Study in Healthy Volunteers and Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allyx Therapeutics (Industry)
Collaborators: Yale University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: ALX-923-102; R01AG073177 (NIH)
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Synapses; Cognition; Neuroprotection; Neurons; mGluR5
MeSH Terms: conditions — Alzheimer Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo capsules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- 50 mg active (Experimental): BMS-984923 50 mg in healthy participants
  Interventions: Drug: BMS-984923
- 50 mg Placebo (Placebo Comparator): Placebo 50 mg in healthy participants
  Interventions: Drug: Placebo
- 100 mg Active (Experimental): BMS-984923 100 mg in healthy participants
  Interventions: Drug: BMS-984923
- 100 mg Placebo (Placebo Comparator): Placebo 100 mg in healthy participants
  Interventions: Drug: Placebo
- 100 mg Active 20d (Experimental): BMS-984923 100 mg in healthy participants 20 days
  Interventions: Drug: BMS-984923
- 100 mg Placebo 20d (Placebo Comparator): Placebo 100 mg in healthy participants 20 days
  Interventions: Drug: Placebo
- 150 mg Active 20d (Experimental): BMS-984923 150 mg in healthy participants 20 days
  Interventions: Drug: BMS-984923
- 150 mg Placebo 20d (Placebo Comparator): Placebo 150 mg in healthy participants 20 days
  Interventions: Drug: Placebo
- 50 mg Active-AD (Experimental): BMS-984923 50 mg
  Interventions: Drug: BMS-984923
- 100 mg Active-AD (Experimental): BMS-984923 100 mg
  Interventions: Drug: BMS-984923
- Placebo-AD (Placebo Comparator): Placebo matching
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-984923 — Capsules
  Other Names: Active
  Arms: 100 mg Active; 100 mg Active 20d; 100 mg Active-AD; 150 mg Active 20d; 50 mg Active-AD; 50 mg active
Drug: Placebo — Capsules
  Other Names: Inactive
  Arms: 100 mg Placebo; 100 mg Placebo 20d; 150 mg Placebo 20d; 50 mg Placebo; Placebo-AD

SUMMARY:
A Phase 1b Multiple Ascending Dose Study of the Safety and Tolerability of BMS-984923 in Healthy Older Adults and Patients with Alzheimer's Disease

DETAILED DESCRIPTION:
This double-blind placebo-controlled study will be completed in 2 stages. The first stage will evaluate 10-days of BID dosing in four ascending dose cohorts in healthy older adults and Stage 2 will examine BMS-984923 dosed BID for 28 days at two dose levels in comparison to Placebo in participants with early AD.

This research study will assess the safety and tolerability of multiple doses of BMS-984923 for the treatment of early Alzheimer's Disease (AD) and investigate the use of synaptic density, measured with positron emission tomography (PET), as an early marker of therapeutic response to treatments that target synapse restoration.

ELIGIBILITY:
Inclusion Criteria Stage 1:

1. Men or women between the ages of 50 and 80 years, inclusive
2. No history of cognitive impairment
3. Capable of providing written informed consent and willing to comply with all study requirements and procedures
4. Participant is not pregnant, lactating, or of childbearing potential

   1. Non-childbearing potential for women is defined as postmenopausal (last natural menses greater than 24 months prior; menopausal status will be documented with serum follicle-stimulating hormone (FSH) or documentation of bilateral tubal ligation or hysterectomy
   2. Male participants who are sexually active with a woman of childbearing potential must agree to use condoms during the trial and for 3 months after the last dose unless the woman is using an acceptable means of birth control. Acceptable forms of birth control include abstinence, birth control pills, or any double combination of intrauterine device (IUD), male or female condom, diaphragm, sponge, and cervical cap.
   3. Male participants must also agree not to donate sperm for 90 days after the last dose.
5. Montreal Cognitive Assessment (MOCA) >25

Exclusion Criteria Stage 1:

1. Body mass index (BMI) >38 kg/m2 or body weight <50 kg.
2. Any significant neurologic disease, such as AD, Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.
3. A current Diagnostic and Statistical Manual of Mental Disorders, Fifth revision (DSM V) diagnosis of active major depression, schizophrenia or bipolar disorder. Participants with depressive symptoms successfully managed by a stable dose of an antidepressant are allowed entry.
4. Positive urine drug screen for amphetamines, barbiturates, benzodiazepines, cocaine, opiates, tetrahydrocannabinol (THC), ethanol or cotinine (stable prescribed amphetamines or benzodiazepines for a non-exclusionary medical condition are permitted) or positive alcohol breathalyzer test
5. Current nicotine use or positive urine cotinine test.
6. History of alcohol or substance abuse or dependence within the past 2 years (DSM IV criteria).
7. Clinically significant or unstable medical condition, including uncontrolled hypertension, uncontrolled diabetes, or significant cardiac, pulmonary, renal, hepatic, endocrine, or other systemic disease in the opinion of the PI, may either put the participant at risk because of participation in the study, or influence the results, or the participant's ability to participate in the study.
8. Any disorder that could interfere with the absorption, distribution, metabolism or excretion of drugs (e.g., small bowel disease, Crohn's disease, celiac disease, or liver disease.)
9. Seropositive for human immunodeficiency virus (HIV).
10. History of acute/chronic hepatitis B or C and/or carriers of hepatitis B (seropositive for hepatitis B surface antigen [HbsAg] or anti-hepatitis C [HCV] antibody).
11. Use of psychoactive medications (typical neuroleptics, narcotic analgesics, antiparkinsonian medications, systemic corticosteroids, or medications with significant central anticholinergic activity) within 2 weeks or 5 half-lives (whichever is greater) prior to study drug administration and for the duration of the trial.
12. Use of medications with potential drug-drug interactions (see Appendix A for a list of these medications) within 2 weeks or 5 half-lives (whichever is greater) prior to study drug administration and for the duration of the trial.
13. Use of anticoagulants within 30 days or 5 half-lives (whichever is greater) prior to study drug administration and for the duration of the trial.
14. Use of another investigational agent within 30 days or 5 half-lives (whichever is greater) prior to screening and for the duration of the trial.
15. Neutropenia defined as absolute neutrophils count of <1,500/microliter.
16. Thrombocytopenia defined as platelet count <100,000/microliter.
17. Clinically significant abnormalities in screening laboratories, including aspartate aminotransferase (AST) >1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) >1.5 times ULN; total bilirubin >1.5 times ULN; serum creatinine >2.0 times ULN.
18. Geriatric Depression Scale (GDS) score of ≥5 and symptoms consistent with a current episode of major depression.

Inclusion Criteria Stage 2

1. Men or women between the ages of 50 and 85 years, inclusive, at the time of first dose of investigational product (IP).
2. Diagnosis of either amnestic mild cognitive impairment (aMCI) or mild dementia due to AD as defined by

   * Mild dementia due to AD

     * National Institute on Aging (NIA)-Alzheimer's Association core clinical criteria for dementia due to probable AD (McKhann 2011) and,
     * Mini Mental Status Exam (MMSE) score between 18 and 26 (inclusive)
     * Clinical Dementia Rating (CDR) global score of 0.5 or 1
   * aMCI due to AD

     * Subjective memory complaint preferably corroborated by an informant and,
     * Normal activities of daily living
     * CDR global score of 0.5
     * aMCI (Petersen 2004) as evidenced by abnormal memory function documented by scoring 1.5 SD below the education adjusted cutoff on the Logical Memory II subscale (Delayed Paragraph Recall) from the Wechsler Memory Scale - Revised (the maximum score is 25), and

       * 8 for 16 or more years of education
       * 4 for 8 15 years of education
       * 2 for 0 7 years of education
3. Stable pharmacological treatment of any other chronic conditions for at least 4 weeks prior to baseline.
4. Neuroimaging (MRI) obtained during screening consistent with the clinical diagnosis of AD as defined in Criteria 2 and without findings of significant exclusionary abnormalities (see Section 6.2.2, exclusion criteria, Number 4).
5. Study partner is available who has frequent contact with the participant (e.g., average of 10 hours per week or more), and can participate in all study partner assessments for the duration of the protocol.
6. Generally healthy with mobility (ambulatory or ambulatory-aided, i.e., walker or cane), vision and hearing (hearing aid permissible) sufficient for compliance with testing procedures as determined by the PI.
7. Must be able to complete all screening evaluations
8. Living at home or in the community (assisted living acceptable)
9. Ability to swallow study medication.
10. Modified Hachinski score ≤4
11. Capable of providing written informed consent and willing to comply with all study requirements and procedures
12. Participant is not pregnant, lactating, or of childbearing potential

    * Non-childbearing potential for women is defined as postmenopausal (last natural menses greater than 24 months prior; menopausal status will be documented with serum FSH or documentation of bilateral tubal ligation or hysterectomy
    * Male participants who are sexually active with a woman of childbearing potential must agree to use condoms during the trial and for 3 months after the last dose unless the woman is using an acceptable means of birth control. Acceptable forms of birth control include abstinence, birth control pills, or any double combination of IUD, male or female condom, diaphragm, sponge, and cervical cap.
    * Male participants must also agree not to donate sperm for 90 days after the last dose.

Exclusion Criteria Stage 2

1. Hospitalization or change of chronic concomitant medication within 4 weeks prior to baseline
2. BMI >38 kg/m2 or body weight <50 kg
3. Any contraindications for MRI studies, such as claustrophobia, the presence of metal (ferromagnetic) implants, metal fragments or foreign objects in the eyes, skin, or body or a cardiac pacemaker.
4. Living in a continuous care nursing facility
5. Screening MRI of the brain indicative of significant abnormality, including, but not limited to, prior hemorrhage or infarct >1 cm3, >3 lacunar infarcts, cerebral contusion, encephalomalacia, aneurysm, vascular malformation, subdural hematoma, hydrocephalus, or space-occupying lesion (e.g., abscess or brain tumor such as meningioma)
6. Clinical or laboratory findings consistent with:

   * Other primary neurodegenerative disease or cognitive disorder (Lewy body disease, frontotemporal lobar disease, Huntington's disease, Jacob-Creutzfeld Disease, Down's syndrome, Parkinson's disease, amyotrophic lateral sclerosis, etc.)
   * Seizure disorder
   * Other infectious, metabolic or systemic diseases affecting the central nervous system (syphilis, present hypothyroidism, present vitamin B12 deficiency, other laboratory abnormalities, etc.)
7. A current DSM V diagnosis of active major depression, schizophrenia or bipolar disorder. Participants with depressive symptoms successfully managed by a stable dose of an antidepressant are allowed entry.
8. Clinically significant or unstable medical condition, including uncontrolled hypertension, uncontrolled diabetes, or significant cardiac, pulmonary, renal, hepatic, endocrine, or other systemic disease that in the opinion of the PI, may either put the participant at risk because of participation in the study, or influence the results, or impair the participant's ability to participate in the study.
9. Disability that may prevent the participant from completing all study requirements (e.g., blindness, deafness, severe language difficulty, etc.)
10. Any disorder that could interfere with the absorption, distribution, metabolism or excretion of drugs (e.g., small bowel disease, Crohn's disease, celiac disease, or liver disease.)
11. Nootropic drugs except stable AD meds (acetylcholinesterase inhibitors and memantine) for 12 weeks prior to baseline
12. History of alcohol or substance abuse or dependence within the past 2 years (DSM IV criteria).
13. Suspected or known allergy to any components of the study treatments
14. Any condition, which in the opinion of the investigator or Project Director (PD) makes the participant unsuitable for inclusion
15. Clinically significant abnormalities in B12 or thyroid function tests (TFTs) that might interfere with the study
16. Use of psychoactive medications (typical neuroleptics, narcotic analgesics, antiparkinsonian medications, systemic corticosteroids, or medications with significant central anticholinergic activity) within 2 weeks or 5 half-lives (whichever is greater) prior to study drug administration and for the duration of the trial
17. Use of medications with potential drug-drug interactions (see Appendix A for a list of these medications) within 2 weeks or 5 half-lives (whichever is greater) prior to study drug administration and for the duration of the trial.
18. Use of anticoagulants within 30 days or 5 half-lives (whichever is greater) prior to study drug administration and for the duration of the trial
19. Use of investigational amyloid lowering therapies within 2 months prior to study drug administration and for the duration of the trial.
20. Use of another investigational agent within 30 days or 5 half-lives (whichever is greater) prior to screening and for the duration of the trial
21. Neutropenia defined as absolute neutrophils count of <1,500/microliter
22. Thrombocytopenia defined as platelet count <100,000/microliter.
23. Clinically significant abnormalities in screening laboratories, including AST >1.5 times ULN; ALT >1.5 times ULN; total bilirubin >1.5 times ULN; serum creatinine >2.0 times ULN
24. GDS score of ≥5 and symptoms consistent with a current episode of major depression.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Stage 1 and Stage 2 Incidence of treatment-emergent adverse events (TEAEs) | Up to 10 days after last dose
  Safety
Stage 1 and Stage 2 Incidence of clinically significant lab abnormalities | Up to 10 days after last dose
  Safety
Stage 1 Incidence of clinically significant changes in safety assessments | Up to 10 days after last dose
  Vital signs, physical exam, electrocardiogram [ECG], Neuropsychiatric Inventory-Questionnaire [NPI Q], Geriatric Depression Scale [GDS], Glasgow Coma Scale [GCS], Montreal Cognitive Assessment [MOCA])
Stage 2 Incidence of clinically significant changes in safety assessments | Up to 10 days after last dose
  Vital signs, physical exam, ECG, NPI Q, GDS, MOCA, and Functional Assessment Questionnaire [FAQ])

SECONDARY OUTCOMES:
Stage 1 and Stage 2 Trough plasma drug concentration at steady state | Up to 10 days after last dose
  plasma concentration as determined by pharmacokinetic modeling
Stage 1 and Stage 2 Area under the curve for the first 24 hours of dosing (AUC24h) and at steady state as determined by PK modeling | Up to 10 days after last dose
  Total plasma concentration as determined by pharmacokinetic modeling
Stage 2 Change from baseline in synaptic density PET | Up to 24 hours after last dose
  Pharmacodynamics
Stage 2 Change from baseline in Alzheimer's Disease Assessment Scale-Cognitive subscale 14 Score range of 0-90, with higher scores indicating greater cognitive impairment. | Up to 7 days after the last dose
  Assessment of cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Mecca, MD, PhD, Study Director — Yale University; Stephanie Post, MD, Principal Investigator — Spaulding Clinical Research (Stage 1); Adam Mecca, MD, PhD, Principal Investigator — Yale University (Stage 2)
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Spaulding Clinical Research, West Bend, Wisconsin

REFERENCES:
- [Background] Haas LT, Salazar SV, Smith LM, Zhao HR, Cox TO, Herber CS, Degnan AP, Balakrishnan A, Macor JE, Albright CF, Strittmatter SM. Silent Allosteric Modulation of mGluR5 Maintains Glutamate Signaling while Rescuing Alzheimer's Mouse Phenotypes. Cell Rep. 2017 Jul 5;20(1):76-88. doi: 10.1016/j.celrep.2017.06.023. PMID 28683325
- [Background] Spurrier J, Nicholson L, Fang XT, Stoner AJ, Toyonaga T, Holden D, Siegert TR, Laird W, Allnutt MA, Chiasseu M, Brody AH, Takahashi H, Nies SH, Perez-Canamas A, Sadasivam P, Lee S, Li S, Zhang L, Huang YH, Carson RE, Cai Z, Strittmatter SM. Reversal of synapse loss in Alzheimer mouse models by targeting mGluR5 to prevent synaptic tagging by C1Q. Sci Transl Med. 2022 Jun;14(647):eabi8593. doi: 10.1126/scitranslmed.abi8593. Epub 2022 Jun 1. PMID 35648810